CLINICAL TRIAL: NCT01095094
Title: Phase II Trial of Ritonavir/Lopinavir in Patients With Progressive of Recurrent High-Grade Gliomas
Brief Title: Ritonavir and Lopinavir in Treating Patients With Progressive or Recurrent High-Grade Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not meet its primary objective
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2307; NCI-2009-01288 (Other: NCI/CTRP); NCT00792987 (obsolete NCT alias)
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-04

CONDITIONS: Brain Tumor; Anaplastic Astrocytoma; Anaplastic Ependymoma; Anaplastic Oligodendroglioma; Brain Stem Glioma; Giant Cell Glioblastoma; Glioblastoma; Gliosarcoma; Mixed Glioma
Keywords: adult brain tumor; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult brain stem glioma; adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; adult mixed glioma; recurrent adult brain tumor
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma | interventions — Ritonavir; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral ritonavir and lopinavir twice daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ritonavir; Drug: lopinavir

INTERVENTIONS:
Drug: ritonavir — Given orally
  Other Names: Norvir; RIT
Drug: lopinavir — Given orally
  Other Names: ABT-378/r

SUMMARY:
RATIONALE: Ritonavir and lopinavir may stop the growth of gliomas by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. PURPOSE: This phase II trial is studying how well giving ritonavir together with lopinavir works in treating patients with progressive or recurrent high-grade glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To evaluate the 6-month progression-free survival in patients with recurrent or progressive high grade gliomas treated with ritonavir and lopinavir. SECONDARY OBJECTIVES: I. To evaluate the toxicity of ritonavir and lopinavir in this patient population. OUTLINE: Patients receive oral ritonavir and lopinavir twice daily in the absence of disease progression or unacceptable toxicity. After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven high grade glioma (WHO grade 3-4) which is progressive or recurrent following radiation therapy with or without chemotherapy
* Patients with previous low grade glioma who progressed after radiotherapy and chemotherapy and are biopsied and found to have a high grade glioma are eligible
* Patients must have recovered from toxicity of prior therapy - An interval of >= 3 months must have elapsed since the completion of the most recent course of radiation therapy
* Minimum interval since last drug therapy: 2 weeks since last non-cytotoxic therapy; 3 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen; 6 weeks since the completion of a nitrosourea containing chemotherapy regimen
* Patients must have a Karnofsky performance status >= 60% (i.e., must be able to care for himself/herself with the occasional help of others)
* Patients must have normal hematologic, renal, and liver function (i.e., absolute neutrophil count >= 1500/mm^3, platelets >= 100,000/mm^3, HgB > 9 d/dl, creatinine =< 1.5mg/dl, total bilirubin =< 1.5mg/dl, transaminases =< 2.5 times the upper limits of the institutional norm)
* Patients must be able to provide written informed consent
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid contraception - Female patients of child-bearing potential must have a negative pregnancy test
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin of carcinoma in situ of the cervix and breast, adequately treated stage I or II cancer from which the patient is in complete remission
* Patients with other prior malignancies must be disease-free for >= 3 years
* Patients must be maintained on a stable corticosteroid regimen from the time of their baseline scan until the start of treatment
* Patients must have a Mini mental state exam score >= 15

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlines in this protocol with reasonable safety
* Patients who are pregnant or breast-feeding
* Patients receiving concurrent therapy for their tumor (with the exception of steroids)
* HIV positive
* Prior therapy with HIV protease inhibitors
* Concurrent therapy with hepatic enzyme inducing anticonvulsant
* Inability to be followed closely at the Cleveland Clinic
* Patients requiring the use of medication well-known contraindicated for concomitant use with lopinavir/ritonavir: amiodarone, astemizole, bepridil, bupropione, cisapride, clorazepate, clozapim, diazepam, encainide, flecainide, flurazepam, meperidine, midazolam, primozide, piroxicam, propafenone, propoxifeno, quinidine, rifabutin, terfenadine, triazolam, zolpidem, dihydroergotamine, ergotamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from medical clinic May 2008 to May 2009.
Groups:
- Arm I: Patients receive oral ritonavir and lopinavir twice daily in the absence of disease progression or unacceptable toxicity.
  ritonavir : Given orally
  lopinavir : Given orally
Period: Overall Study
Arm/Group | Arm I
Started | 19
Completed | 16
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 19
Age, Customized [Number; unit: Participants]
  30-39 years | 4
  40-49 years | 5
  50-59 years | 7
  60-69 years | 1
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Number of patients that remained disease free at 6 months from start of treatment.
Time Frame: At 6 months
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 16
participants | 4

2. Secondary Outcome: Grade 3-5 Toxicity as Assessed by NCI CTC v3.0
Description: Number of participants with adverse events grades 3-5. For a detailed list of adverse events see the adverse event module.
Time Frame: at 6 months from start of treatment
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 19
participants | 7

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected on all patients while on study over a 3 year 5 month period.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 5/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=19)
Vomiting (Gastrointestinal disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Incontinence, urinary (Renal and urinary disorders) | 1
Edema: limb (General disorders) | 1
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=19)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Elevated AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1
Ataxia (Nervous system disorders) | 1
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 5
Cognitive disturbance (Nervous system disorders) | 2
Confusion (Nervous system disorders) | 2
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 4
Edema: limb (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7
Flu-like syndrome (General disorders) | 1
Bad Breath (Gastrointestinal disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
hot Flashes/Flushes (Endocrine disorders) | 1
Incontinence, urinary (Renal and urinary disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Memory impairment (Nervous system disorders) | 4
Mood alteration - Anxiety (Nervous system disorders) | 1
Mood alteration - Depression (Psychiatric disorders) | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 4
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Neuropathy: cranial - CN XII Motor-tongue (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 1
Ocular/Visual - Other (Specify, Foggy Vision) (Eye disorders) | 2
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain - Head/headache (Nervous system disorders) | 3
Thrombocytopenia (Investigations) | 3
Potassium, serum-low (hypokalemia) (Investigations) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Rigors/chills (General disorders) | 1
Salivary gland changes/ increased saliva (Gastrointestinal disorders) | 2
Seizure (Nervous system disorders) | 3
Somnolence/depressed level of consciousness (Nervous system disorders) | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 4
Sweating (diaphoresis) (General disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 7
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight Loss (Investigations) | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes